CLINICAL TRIAL: NCT05447637
Title: A Multi-center Prospective Observational Study of Community Urology Practices Applying Germline Genetic Testing for Prostate Cancer Patients (PROCLAIM)
Brief Title: PROCLAIM: Germline Genetic Testing for Prostate Cancer Patients
Status: Completed | Type: Observational
Sponsor: Invitae Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: INVPC-1000
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: None Retained — Blood samples provided for clinical genetic testing that include DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals who meet NCCN Testing Criteria
  Interventions: Diagnostic Test: Invitae multi-cancer gene panel
- Individuals who do not meet NCCN Testing Criteria
  Interventions: Diagnostic Test: Invitae multi-cancer gene panel

INTERVENTIONS:
Diagnostic Test: Invitae multi-cancer gene panel — Invitae's multi-cancer panel tests for 84 genes associated with hereditary cancer risk.

SUMMARY:
This registry is for men who have prostate cancer and have had multigene panel hereditary testing. The registry will gather data on genetic testing results and how that information may change physician treatment or follow up recommendations. It will also gather data on the patient's experience with genetic testing, through a post-test survey to be completed 60-90days after results have been received and discussed with their provider.

DETAILED DESCRIPTION:
This registry will enroll men with prostate cancer who have done multi-gene testing for their cancer. Patients will be enrolled into two cohorts, one for individuals who meet current NCCN testing guidelines, and one for individuals who do not meet current NCCN guidelines.

The main goal of this Registry is to assess whether nationally developed guidelines used to select patients for hereditary testing are adequate to identify all patients with prostate cancer who may benefit from testing. Patients will completed a post-test survey regarding their testing experience and clinicians will be asked to provide additional medical records review information via the Clinician Report Form.

ELIGIBILITY:
Inclusion Criteria:

* Men ages 18-90 who have been prescribed genetic testing as part of their clinical care
* Have prostate cancer at any stage, either actively under treatment or being followed who either: 1. meet NCCN criteria for testing or 2. do not meet NCCN criteria for testing
* Patients who are naive to clinical genetic testing for BRCA1/BRCA2 (single gene panel testing)

Exclusion Criteria:

* Mental or cognitive impairment that interferes with ability to provide informed consent

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men
Study Population: Men who have a diagnosis of prostate cancer who have not previously undergone testing for multi-gene hereditary cancer risk.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of pathogenic and likely pathogenic genes in the patient population | to be assessed at baseline only
  Identify the diagnostic yield of pathogenic/likely pathogenic variants in known cancer syndrome genes in patients with prostate cancer, using the Invitae 84 gene multi-cancer panel. These rates will be compared between the two cohorts.

SECONDARY OUTCOMES:
Evaluate the sensitivity of current NCCN criteria for germline genetic testing for identifying prostate cancer patients that have pathogenic/likely pathogenic variants | at baseline only
  Compare rates of pathogenic / likely pathogenic variants found in both cohorts after testing using the Invitae 84 gene multi cancer panel.
Evaluate the impact of genetic test results on clinical management decisions | 60-90 days post test results received.
  Post-Test surveys for patients and the clinician report form will assess whether changes to clinical management were made as a result of the test results.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Genesis Healthcare Partners, San Diego, California
  - Invitae, San Francisco, California
  - Department of Bioengineering and Therapeutic Sciences, University of California San Francisco, San Francisco, California
  - Volunteer Faculty, University of California San Francisco, San Francisco, California
  - Colorado Urology, Lakewood, Colorado
  - Advanced Urology Institute, St. Petersburg, Florida
  - Florida Urology Partners, Tampa, Florida
  - TGH Cancer Institute, Tampa, Florida
  - North Georgia Urology, Dalton, Georgia
  - Associated Urological Specialists, Chicago Ridge, Illinois
  - University Urology Associates of New Jersey, Hamilton, New Jersey
  - Perlmutter Cancer Center, NYU Langone Health, New York, New York, New York
  - Associated Medical Professionals, Syracuse, New York
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - Urology Partners, Arlington, Texas
  - Urology Austin, Austin, Texas
  - Urosurgery Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD at this time.